CLINICAL TRIAL: NCT06450327
Title: Resistant Hypertension An Open, Complicated ("Cum Plicare") or Complex ("Cum Plexus")
Brief Title: Resistant Hypertension An Open, Complicated ("Cum Plicare") or Complex ("Cum Plexus") Syndrome?
Status: Recruiting | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Tatiane De Azevedo Rubio, Principal Investigator, University of Campinas, Brazil
Other Study IDs: 57573922.0.0000.5415
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Hypertension; Resistant Hypertension
Keywords: autonomic nervous system; resistant hypertension; arterial hypertension; refractory hypertension; baroreceptors
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normotensives - apparently healthy: Group of non-hypertensive participants
  Interventions: Other: This is a cross-sectional observational study
- Controlled hypertension: Participants diagnosed with primary arterial hypertension and undergoing outpatient follow-up
  Interventions: Other: This is a cross-sectional observational study
- Resistant Hypertension: Participants diagnosed with primary arterial hypertension using 3 or more antihypertensive medications, one of which is preferably a thiazide diuretic
  Interventions: Other: This is a cross-sectional observational study
- Refractory Hypertension: Participants diagnosed with primary arterial hypertension using 5 or more antihypertensive medications.
  Interventions: Other: This is a cross-sectional observational study

INTERVENTIONS:
Other: This is a cross-sectional observational study — There will be no intervention in the study.

SUMMARY:
Resistant arterial hypertension (RAH) is a complex and multifactorial syndrome, with hyperactivity of the sympathetic nervous system (SNS) and reduction of vagal activity being considered some of the main causes of refractoriness to treatment. Seen from the outside, it resembles a complicated (see lat. "Cum plicate") or complex disease (see lat. "Cum plexus"), Chaotic with the participation of several open systems. For example, in recent years some relationships have been demonstrated between the autonomic nervous systems, synaptic mediators, hormones, inflammatory and immune responses. However, these findings have not been investigated together and systematically. In the present project, we intend to establish and compare, in an integrated way, the clinical alterations present in RAH (resistant and refractory), hemodynamic variables, autonomous activity (sympathetic and baroreflex) and interactions with the neuroimmune-endocrine systems. To this end, we will test the hypothesis that resistant patients have greater damage to the autonomic nervous system (ANS) associated with exacerbated systemic and hormonal inflammatory profile, including SNA mediators (noradrenaline and acetylcholinesterase). This is also intended to determine the behavior (deterministic or chaotic) of the systems evaluated (mentioned above) in volunteers with RAH. Sample and methods: The sample space (calculated) will consist of 72 individuals, being: - 18 refractory hypertensive (HRT); II- 18 resistant hypertensive patients (HRfT); III- 18 controlled hypertensive (1-2 drugs) (CAH); and IV- 18 healthy normotensive individuals. This is a prospective, double-blind study (patient and professional-technician), paired (1 X 4), in which the 72 volunteers will be evaluated by the methods set out below. We will also have the chance to observe whether resistant and refractory hypertension share the same pathophysiological bases and clinical manifestations ("deterministic-isolated or cardiovascular chaos") by analyzing the patterns of cardiovascular variability (MAPA and Holter) (SpaceLabs, USA; DynaMap, Brazil), inflammatory and hormonal mediators (ELISA) in the resistant hypertension - RHT and refratary hypertension - HfRT groups. Central pressure (CP) and arterial stiffness (pulse wave velocity, VOP) (Sphymocor, ATCor, USA) will also be assessed. Healthy normotensive (NT) and controlled hypertension (CAH) will be evaluated in an identical way to control the other groups. Perspectives: The findings will improve the clinical knowledge based on pathophysiology about Resistant Hypertension and, mainly, the bases of pharmacological treatment and with implantable devices (stimulation of baroreceptors and sympathetic denervation) used in this condition.

DETAILED DESCRIPTION:
Cardiovascular Autonomic Modulation Procedures for spectral analysis of pulse interval (heart rate variability) and systolic blood pressure variability have been described in the literature41-44. Each heartbeat will be identified using a specialized algorithm implemented in Matlab MT software (MATLAB 6.0, Mathworks, USA ) and which automatically detects PAS and PAD waves. The pulse interval or R-R interval will be calculated as the difference between the start and end points of the cycle (t1-t0). The power spectral density of the PAS and R-R interval will be calculated using the Fast Fourier Transform and the Welch method over 16,384 points with a Hanning window and 50% overlap. The spectral bands evaluated for humans were defined according to literature references: very low frequency (MBF: 0.007-0.04Hz), low frequency (BF: 0.04-0.15Hz), high frequency (AF: 0. 15-0.4 Hz) and full power [130]. Baroreflex sensitivity will be inferred from the alpha index (HR BF ratio in ms2 / SBP BF ratio in mmHg).

ABPM - It will be performed with the CardioMAPA Monitor - Cardios - Brazil, with standardized measurements every 15 minutes during the waking period, and every 20 minutes during the sleeping period. The data will be considered valid when monitoring takes place for a minimum period of 21 hours with a minimum number of forty measurements during wakefulness and ten measurements during sleep.

Determination of Central Blood Pressure and Amplification Index (AIx) - The SphygmoCor CPV system (AtCor Medical, USA) is a sophisticated non-invasive diagnostic tool for clinical assessment of central blood pressure. This system derives central aortic pulse wave pressure (systolic, diastolic, and pulse) using pulse wave pressure recorded by the radial artery. Pulse wave analysis predicts parameters including PAC and indications of vascular stiffness. Measurements are made using a pressure transducer (tonometer) positioned in the required artery and then the pulse wave is recorded. Furthermore, this equipment provides information on arterial stiffness by analyzing the Augmentation Index [Amplification Index (AIx)], defined by the ratio between the pressure determined by the reflected wave and the ejection wave capable of providing information on arterial stiffness.

Assessment of Clinical Parameters - BP measurements will be taken according to the recommendations recommended by the VIII Brazilian Guidelines on Arterial Hypertension using a digital sphygmomanometer (Omron HEM-711DLX). Pulse pressure (PP) will be calculated from the difference between SBP and DBP values. All individuals will undergo ambulatory BP monitoring (ABPM) for a period of 24 hours using the Spacelabs 90217 equipment (Spacelabs Inc, Redmon, WA, USA). Patients will be instructed to maintain and record normal daily activities. The averages of SBP, DBP and PP will be evaluated.

Assessment of Biochemical and Inflammatory Parameters - Fasting blood samples will be collected and the following tests will be carried out: glucose, glycated hemoglobin A1C, total cholesterol and fractions, urea, creatinine, renin, aldosterone, cortisol, creatinine clearance and microalbuminuria. The biomarkers norepinephrine, dopamine, adrenaline, adrenocorticotropic hormones (ACTH) and cortisol, acetylcholinesterase, ultrasensitive C-reactive protein, interleukins 2, 8, 10 and 12 (IL-2, IL-8, IL-10 and IL-12) will be determined by ELISA according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 35 years of age diagnosed with resistant arterial hypertension (RH), in accordance with the latest international and national guidelines;
* be able to understand, verbalize and answer questions;
* agree to participate in the study and sign the Informed Consent Form;
* after clearly understanding it;
* be under regular follow-up at the UNICAMP Cardiovascular Pharmacology outpatient clinic for at least six months;
* have proven adherence to non-pharmacological and pharmacological treatment;
* women in the reproductive phase must be using a proven effective contraceptive method.

Exclusion Criteria:

* clinical history or clinical symptoms of heart failure;
* patients with dilated cardiomyopathies, valvular heart disease, pericardial disorders;
* patients with cerebrovascular disease or peripheral arterial disease, nephropathies, liver diseases, smoking, autoimmune diseases and use of illicit substances;
* any abnormal condition that may interfere with the results of the study or the health of the volunteer, as judged by the researcher;
* women who are pregnant or intend to become pregnant;
* current participation in another investigative study;
* major depression or other relevant psychiatric disorders.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the Resistant Hypertension Outpatient Clinic of the HC of UNICAMP and FAMERP - Faculty of Medicine of São José do Rio Preto. During the first six months of follow-up, ambulatory BP monitoring (ABPM) and optimization of pharmacological therapy will be carried out, including strict control of treatment adherence (pill count) and dietary guidelines. Furthermore, possible causes of secondary hypertension will be investigated and excluded.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 4 weeks
  through MAPA using non-linear calculations from Chaos Theory
Heart Rate | 4 weeks
  through MAPA using non-linear calculations from Chaos Theory
Level of TNF-α | 10 weeks
  Analysis of inflammatory responses associated with blood pressure variability
Level of IL1β, IL-6 | 10 weeks
  Analysis of inflammatory responses associated with blood pressure variability

CONTACTS AND LOCATIONS:
Locations (1):
- Tatiane de Azevedo Rubio, Votuporanga, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
There will be no data sharing.

REFERENCES:
- [Background] Carey RM, Calhoun DA, Bakris GL, Brook RD, Daugherty SL, Dennison-Himmelfarb CR, Egan BM, Flack JM, Gidding SS, Judd E, Lackland DT, Laffer CL, Newton-Cheh C, Smith SM, Taler SJ, Textor SC, Turan TN, White WB; American Heart Association Professional/Public Education and Publications Committee of the Council on Hypertension; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Genomic and Precision Medicine; Council on Peripheral Vascular Disease; Council on Quality of Care and Outcomes Research; and Stroke Council. Resistant Hypertension: Detection, Evaluation, and Management: A Scientific Statement From the American Heart Association. Hypertension. 2018 Nov;72(5):e53-e90. doi: 10.1161/HYP.0000000000000084. PMID 30354828
- [Background] Persell SD. Prevalence of resistant hypertension in the United States, 2003-2008. Hypertension. 2011 Jun;57(6):1076-80. doi: 10.1161/HYPERTENSIONAHA.111.170308. Epub 2011 Apr 18. PMID 21502568
- [Background] Modolo R, de Faria AP, Sabbatini AR, Barbaro NR, Ritter AM, Moreno H. Refractory and resistant hypertension: characteristics and differences observed in a specialized clinic. J Am Soc Hypertens. 2015 May;9(5):397-402. doi: 10.1016/j.jash.2015.03.005. Epub 2015 Mar 19. PMID 25979412
- [Background] Modolo R, de Faria AP, Almeida A, Moreno H. Resistant or refractory hypertension: are they different? Curr Hypertens Rep. 2014 Oct;16(10):485. doi: 10.1007/s11906-014-0485-1. PMID 25139782
- [Background] Gaddam KK, Nishizaka MK, Pratt-Ubunama MN, Pimenta E, Aban I, Oparil S, Calhoun DA. Characterization of resistant hypertension: association between resistant hypertension, aldosterone, and persistent intravascular volume expansion. Arch Intern Med. 2008 Jun 9;168(11):1159-64. doi: 10.1001/archinte.168.11.1159. PMID 18541823
- [Background] Martins LC, Figueiredo VN, Quinaglia T, Boer-Martins L, Yugar-Toledo JC, Martin JF, Demacq C, Pimenta E, Calhoun DA, Moreno H Jr. Characteristics of resistant hypertension: ageing, body mass index, hyperaldosteronism, cardiac hypertrophy and vascular stiffness. J Hum Hypertens. 2011 Sep;25(9):532-8. doi: 10.1038/jhh.2010.95. Epub 2010 Oct 7. PMID 20927128
- [Background] Figueiredo VN, Yugar-Toledo JC, Martins LC, Martins LB, de Faria AP, de Haro Moraes C, Sierra C, Coca A, Moreno H. Vascular stiffness and endothelial dysfunction: Correlations at different levels of blood pressure. Blood Press. 2012 Feb;21(1):31-8. doi: 10.3109/08037051.2011.617045. Epub 2011 Oct 27. PMID 22029740
- [Background] de Faria AP, Modolo R, Fontana V, Moreno H. Adipokines: novel players in resistant hypertension. J Clin Hypertens (Greenwich). 2014 Oct;16(10):754-9. doi: 10.1111/jch.12399. Epub 2014 Sep 4. PMID 25186286
- [Background] Barbaro NR, de Araujo TM, Tanus-Santos JE, Anhe GF, Fontana V, Moreno H. Vascular Damage in Resistant Hypertension: TNF-Alpha Inhibition Effects on Endothelial Cells. Biomed Res Int. 2015;2015:631594. doi: 10.1155/2015/631594. Epub 2015 Oct 4. PMID 26504819
- [Background] Barbaro NR, Fontana V, Modolo R, De Faria AP, Sabbatini AR, Fonseca FH, Anhe GF, Moreno H. Increased arterial stiffness in resistant hypertension is associated with inflammatory biomarkers. Blood Press. 2015 Feb;24(1):7-13. doi: 10.3109/08037051.2014.940710. Epub 2014 Jul 25. PMID 25061978
- [Background] Dudenbostel T, Siddiqui M, Oparil S, Calhoun DA. Refractory Hypertension: A Novel Phenotype of Antihypertensive Treatment Failure. Hypertension. 2016 Jun;67(6):1085-92. doi: 10.1161/HYPERTENSIONAHA.116.06587. Epub 2016 Apr 18. No abstract available. PMID 27091893
- [Background] Acelajado MC, Hughes ZH, Oparil S, Calhoun DA. Treatment of Resistant and Refractory Hypertension. Circ Res. 2019 Mar 29;124(7):1061-1070. doi: 10.1161/CIRCRESAHA.118.312156. PMID 30920924
- [Background] Acelajado MC, Pimenta E, Calhoun DA. Salt and aldosterone: a concert of bad effects. Hypertension. 2010 Nov;56(5):804-5. doi: 10.1161/HYPERTENSIONAHA.110.160960. Epub 2010 Oct 4. No abstract available. PMID 20921423
- [Background] Ritter AM, de Faria AP, Barbaro N, Sabbatini AR, Correa NB, Brunelli V, Amorim R, Modolo R, Moreno H. Crosstalk between obesity and MMP-9 in cardiac remodelling -a cross-sectional study in apparent treatment-resistant hypertension. Blood Press. 2017 Apr;26(2):122-129. doi: 10.1080/08037051.2016.1249336. Epub 2016 Nov 8. PMID 27825280
- [Background] de Haro Moraes C, Figueiredo VN, de Faria AP, Barbaro NR, Sabbatini AR, Quinaglia T, Ferreira-Melo SE, Martins LC, Demacq C, Junior HM. High-circulating leptin levels are associated with increased blood pressure in uncontrolled resistant hypertension. J Hum Hypertens. 2013 Apr;27(4):225-30. doi: 10.1038/jhh.2012.29. Epub 2012 Jul 19. PMID 22810172
- [Background] Faria AP, Ritter AMV, Gasparetti CS, Correa NB, Brunelli V, Almeida A, Pires NF, Modolo R, Moreno Junior H. A Proposed Inflammatory Score of Circulating Cytokines/Adipokines Associated with Resistant Hypertension, but Dependent on Obesity Parameters. Arq Bras Cardiol. 2019 Apr;112(4):383-389. doi: 10.5935/abc.20190032. Epub 2019 Feb 28. PMID 30843931
- [Background] Ritter AM, Fontana V, Faria AP, Modolo R, Barbaro NR, Sabbatini AR, Peres H, Biagi C, Silva PS, Lopes PC, Tanus-Santos JE, Coelho EB, Moreno H. Association of Mineralocorticoid Receptor Polymorphism I180V With Left Ventricular Hypertrophy in Resistant Hypertension. Am J Hypertens. 2016 Feb;29(2):245-50. doi: 10.1093/ajh/hpv070. Epub 2015 Jun 6. PMID 26049084
- [Background] Bisognano JD, Bakris G, Nadim MK, Sanchez L, Kroon AA, Schafer J, de Leeuw PW, Sica DA. Baroreflex activation therapy lowers blood pressure in patients with resistant hypertension: results from the double-blind, randomized, placebo-controlled rheos pivotal trial. J Am Coll Cardiol. 2011 Aug 9;58(7):765-73. doi: 10.1016/j.jacc.2011.06.008. PMID 21816315
- [Background] Dudenbostel T, Acelajado MC, Pisoni R, Li P, Oparil S, Calhoun DA. Refractory Hypertension: Evidence of Heightened Sympathetic Activity as a Cause of Antihypertensive Treatment Failure. Hypertension. 2015 Jul;66(1):126-33. doi: 10.1161/HYPERTENSIONAHA.115.05449. Epub 2015 May 18. PMID 25987662
- [Background] Muxfeldt ES, de Souza F, Margallo VS, Salles GF. Cardiovascular and renal complications in patients with resistant hypertension. Curr Hypertens Rep. 2014 Sep;16(9):471. doi: 10.1007/s11906-014-0471-7. PMID 25079852
- [Background] Muiesan ML, Salvetti M, Rizzoni D, Paini A, Agabiti-Rosei C, Aggiusti C, Agabiti Rosei E. Resistant hypertension and target organ damage. Hypertens Res. 2013 Jun;36(6):485-91. doi: 10.1038/hr.2013.30. Epub 2013 Apr 18. PMID 23595044
- [Background] Metelka R. Heart rate variability--current diagnosis of the cardiac autonomic neuropathy. A review. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2014 Sep;158(3):327-38. doi: 10.5507/bp.2014.025. Epub 2014 Jul 4. PMID 25004914
- [Background] Salles GF, Cardoso CR, Fiszman R, Muxfeldt ES. Prognostic impact of baseline and serial changes in electrocardiographic left ventricular hypertrophy in resistant hypertension. Am Heart J. 2010 May;159(5):833-40. doi: 10.1016/j.ahj.2010.02.012. PMID 20435193
- [Background] Salles GF, Ribeiro FM, Guimaraes GM, Muxfeldt ES, Cardoso CR. A reduced heart rate variability is independently associated with a blunted nocturnal blood pressure fall in patients with resistant hypertension. J Hypertens. 2014 Mar;32(3):644-51. doi: 10.1097/HJH.0000000000000068. PMID 24445393
- [Background] Dudenbostel T, Calhoun DA. Resistant hypertension, obstructive sleep apnoea and aldosterone. J Hum Hypertens. 2012 May;26(5):281-7. doi: 10.1038/jhh.2011.47. Epub 2011 Jun 9. PMID 21654850
- [Background] Muxfeldt ES, Margallo VS, Guimaraes GM, Salles GF. Prevalence and associated factors of obstructive sleep apnea in patients with resistant hypertension. Am J Hypertens. 2014 Aug;27(8):1069-78. doi: 10.1093/ajh/hpu023. Epub 2014 Apr 4. PMID 24705438
- [Background] Agashe S, Petak S. Cardiac Autonomic Neuropathy in Diabetes Mellitus. Methodist Debakey Cardiovasc J. 2018 Oct-Dec;14(4):251-256. doi: 10.14797/mdcj-14-4-251. PMID 30788010
- [Background] Grassi G. Assessment of sympathetic cardiovascular drive in human hypertension: achievements and perspectives. Hypertension. 2009 Oct;54(4):690-7. doi: 10.1161/HYPERTENSIONAHA.108.119883. Epub 2009 Aug 31. PMID 19720958
- [Background] Grassi G, Pisano A, Bolignano D, Seravalle G, D'Arrigo G, Quarti-Trevano F, Mallamaci F, Zoccali C, Mancia G. Sympathetic Nerve Traffic Activation in Essential Hypertension and Its Correlates: Systematic Reviews and Meta-Analyses. Hypertension. 2018 Aug;72(2):483-491. doi: 10.1161/HYPERTENSIONAHA.118.11038. Epub 2018 Jun 18. PMID 29915014
- [Background] Kasiakogias A, Tsioufis C, Dimitriadis K, Konstantinidis D, Koumelli A, Leontsinis I, Andrikou E, Vogiatzakis N, Marinaki S, Petras D, Fragoulis C, Konstantinou K, Papademetriou V, Tousoulis D. Cardiovascular morbidity of severe resistant hypertension among treated uncontrolled hypertensives: a 4-year follow-up study. J Hum Hypertens. 2018 Jul;32(7):487-493. doi: 10.1038/s41371-018-0065-y. Epub 2018 May 1. PMID 29713047
- [Background] Feng YN, Xiao H, Zhang YY. [Research advances of autonomic nervous system in the regulation of cardiac inflammation]. Sheng Li Xue Bao. 2019 Apr 25;71(2):225-234. Chinese. PMID 31008482
- [Background] Palatini P, Dorigatti F, Zaetta V, Mormino P, Mazzer A, Bortolazzi A, D'Este D, Pegoraro F, Milani L, Mos L; HARVEST Study Group. Heart rate as a predictor of development of sustained hypertension in subjects screened for stage 1 hypertension: the HARVEST Study. J Hypertens. 2006 Sep;24(9):1873-80. doi: 10.1097/01.hjh.0000242413.96277.5b. PMID 16915038
- [Background] Li YF, LaCroix C, Freeling J. Specific subtypes of nicotinic cholinergic receptors involved in sympathetic and parasympathetic cardiovascular responses. Neurosci Lett. 2009 Oct 2;462(1):20-3. doi: 10.1016/j.neulet.2009.06.081. Epub 2009 Jun 30. PMID 19573576
- [Background] Bissinger A. Cardiac Autonomic Neuropathy: Why Should Cardiologists Care about That? J Diabetes Res. 2017;2017:5374176. doi: 10.1155/2017/5374176. Epub 2017 Oct 29. PMID 29214181
- [Background] Karakas M, Koenig W. Sympathetic nervous system: a crucial player modulating residual cardiovascular risk. Circ Res. 2013 Jan 4;112(1):13-6. doi: 10.1161/CIRCRESAHA.112.281097. No abstract available. PMID 23287453
- [Background] Shaffer F, McCraty R, Zerr CL. A healthy heart is not a metronome: an integrative review of the heart's anatomy and heart rate variability. Front Psychol. 2014 Sep 30;5:1040. doi: 10.3389/fpsyg.2014.01040. eCollection 2014. PMID 25324790
- [Background] Pierdomenico SD, Lapenna D, Bucci A, Di Tommaso R, Di Mascio R, Manente BM, Caldarella MP, Neri M, Cuccurullo F, Mezzetti A. Cardiovascular outcome in treated hypertensive patients with responder, masked, false resistant, and true resistant hypertension. Am J Hypertens. 2005 Nov;18(11):1422-8. doi: 10.1016/j.amjhyper.2005.05.014. PMID 16280275
- [Background] Rozanski A, Blumenthal JA, Kaplan J. Impact of psychological factors on the pathogenesis of cardiovascular disease and implications for therapy. Circulation. 1999 Apr 27;99(16):2192-217. doi: 10.1161/01.cir.99.16.2192. PMID 10217662
- [Background] Kaye DM, Lefkovits J, Jennings GL, Bergin P, Broughton A, Esler MD. Adverse consequences of high sympathetic nervous activity in the failing human heart. J Am Coll Cardiol. 1995 Nov 1;26(5):1257-63. doi: 10.1016/0735-1097(95)00332-0. PMID 7594040
- [Background] de Souza WA, Yugar-Toledo JC, Bergsten-Mendes G, Sabha M, Moreno H Jr. Effect of pharmaceutical care on blood pressure control and health-related quality of life in patients with resistant hypertension. Am J Health Syst Pharm. 2007 Sep 15;64(18):1955-61. doi: 10.2146/ajhp060547. PMID 17823108
- [Background] Reule S, Drawz PE. Heart rate and blood pressure: any possible implications for management of hypertension? Curr Hypertens Rep. 2012 Dec;14(6):478-84. doi: 10.1007/s11906-012-0306-3. PMID 22972532
- [Background] Dalal J, Dasbiswas A, Sathyamurthy I, Maddury SR, Kerkar P, Bansal S, Thomas J, Mandal SC, Mookerjee S, Natarajan S, Kumar V, Chandra N, Khan A, Vijayakumar R, Sawhney JPS. Heart Rate in Hypertension: Review and Expert Opinion. Int J Hypertens. 2019 Feb 19;2019:2087064. doi: 10.1155/2019/2087064. eCollection 2019. PMID 30915238
- [Background] Martinez PF, Okoshi MP. Heart Rate Variability in Coexisting Diabetes and Hypertension. Arq Bras Cardiol. 2018 Jul;111(1):73-74. doi: 10.5935/abc.20180118. No abstract available. PMID 30110047
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Laurent S, Alivon M, Beaussier H, Boutouyrie P. Aortic stiffness as a tissue biomarker for predicting future cardiovascular events in asymptomatic hypertensive subjects. Ann Med. 2012 Jun;44 Suppl 1:S93-7. doi: 10.3109/07853890.2011.653398. PMID 22713154
- [Background] Pettersen KH, Bugenhagen SM, Nauman J, Beard DA, Omholt SW. Arterial stiffening provides sufficient explanation for primary hypertension. PLoS Comput Biol. 2014 May 22;10(5):e1003634. doi: 10.1371/journal.pcbi.1003634. eCollection 2014 May. PMID 24853828
- [Background] Mitchell GF, Hwang SJ, Vasan RS, Larson MG, Pencina MJ, Hamburg NM, Vita JA, Levy D, Benjamin EJ. Arterial stiffness and cardiovascular events: the Framingham Heart Study. Circulation. 2010 Feb 2;121(4):505-11. doi: 10.1161/CIRCULATIONAHA.109.886655. Epub 2010 Jan 18. PMID 20083680
- [Background] Barroso WKS, Rodrigues CIS, Bortolotto LA, Mota-Gomes MA, Brandao AA, Feitosa ADM, Machado CA, Poli-de-Figueiredo CE, Amodeo C, Mion Junior D, Barbosa ECD, Nobre F, Guimaraes ICB, Vilela-Martin JF, Yugar-Toledo JC, Magalhaes MEC, Neves MFT, Jardim PCBV, Miranda RD, Povoa RMDS, Fuchs SC, Alessi A, Lucena AJG, Avezum A, Sousa ALL, Pio-Abreu A, Sposito AC, Pierin AMG, Paiva AMG, Spinelli ACS, Nogueira ADR, Dinamarco N, Eibel B, Forjaz CLM, Zanini CRO, Souza CB, Souza DDSM, Nilson EAF, Costa EFA, Freitas EV, Duarte EDR, Muxfeldt ES, Lima Junior E, Campana EMG, Cesarino EJ, Marques F, Argenta F, Consolim-Colombo FM, Baptista FS, Almeida FA, Borelli FAO, Fuchs FD, Plavnik FL, Salles GF, Feitosa GS, Silva GVD, Guerra GM, Moreno Junior H, Finimundi HC, Back IC, Oliveira Filho JB, Gemelli JR, Mill JG, Ribeiro JM, Lotaif LAD, Costa LSD, Magalhaes LBNC, Drager LF, Martin LC, Scala LCN, Almeida MQ, Gowdak MMG, Klein MRST, Malachias MVB, Kuschnir MCC, Pinheiro ME, Borba MHE, Moreira Filho O, Passarelli Junior O, Coelho OR, Vitorino PVO, Ribeiro Junior RM, Esporcatte R, Franco R, Pedrosa R, Mulinari RA, Paula RB, Okawa RTP, Rosa RF, Amaral SLD, Ferreira-Filho SR, Kaiser SE, Jardim TSV, Guimaraes V, Koch VH, Oigman W, Nadruz W. Brazilian Guidelines of Hypertension - 2020. Arq Bras Cardiol. 2021 Mar;116(3):516-658. doi: 10.36660/abc.20201238. No abstract available. English, Portuguese. PMID 33909761